CLINICAL TRIAL: NCT05166850
Title: Evidence Based Targeted Water Sanitation, and Hygiene Interventions to Reduce Cholera in Hotspots in the Democratic Republic of the Congo
Brief Title: Preventative Intervention for Cholera for 7 Days
Acronym: PICHA-7
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: University of New Mexico (Other); Wellcome Sanger Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00009848
Record Dates: First submitted 2021-12-08; First posted 2021-12-22 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Cholera; Water-Related Diseases; Diarrhea Infectious
MeSH Terms: conditions — Cholera; Waterborne Diseases; Dysentery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preventive-Intervention-for-Cholera-for-7-Days (PICHA7) Mobile Health (mHealth) Program (Experimental): Preventive-Intervention-for-Cholera-for-7-Days (PICHA7) mHealth program promoting handwashing with soap and water treatment for diarrhea patient households
  Interventions: Behavioral: PICHA7 mHealth program; Other: Standard Arm
- Standard Arm (Active Comparator): Standard recommendation in the Democratic Republic of the Congo for diarrhea patients upon discharge from health facilities
  Interventions: Other: Standard Arm

INTERVENTIONS:
Behavioral: PICHA7 mHealth program — The PICHA7 mHealth program is first delivered during a health facility visit by a health promoter bedside to a diarrhea patient (adults and child) and their accompanying household members during the time of illness followed by two home visits during the 7-day high risk period for diarrheal disease transmission. The health promoter delivers a pictorial WASH module on how diarrhea can spread, and instructions on handwashing with soap, water treatment, and safe water storage. A diarrhea prevention package is provided containing: a one-month supply of chlorine tablets for water treatment, a soapy water bottle for handwashing, a handwashing station, and a water vessel with a lid and tap to ensure safe water storage. After health facility delivery of the program, patient households receive weekly voice and text messages from the PICHA7 mHealth program over 12 months on the recommended WASH behaviors.
  Arms: Preventive-Intervention-for-Cholera-for-7-Days (PICHA7) Mobile Health (mHealth) Program
Other: Standard Arm — Standard message given in the Democratic Republic of the Congo to diarrhea patients at health facility discharge on use of oral rehydration solution

SUMMARY:
The first objective of our study is to develop a theory-driven evidence-based targeted water, sanitation, and hygiene (WASH) intervention for household members of diarrhea patients in South Kivu, Democratic Republic of the Congo (DRC) through formative research and community engagement. The second objective is to conduct a randomized controlled trial of 2,320 household members of 580 severe diarrhea patients to evaluate the effectiveness of the developed targeted WASH intervention in terms of: 1. reducing diarrheal diseases household members of cholera and severe diarrhea patients; and 2. increasing WASH behaviors.

DETAILED DESCRIPTION:
This study develops and evaluates a targeted water, sanitation, and hygiene (WASH) intervention to reduce cholera and severe diarrhea among the household members of diarrhea patients in South Kivu, Democratic Republic of the Congo (DRC) through formative research and a randomized controlled trial. This study will also investigate cholera and severe diarrhea transmission dynamics among diarrhea patient households using genomics and a risk factor analysis. The study will be divided into two phases: (1) the Formative Research and Intervention Development Phase; and (2) the Intervention Implementation and Evaluation Phase.

In the two arm randomized controlled trial of diarrhea patient households, we compare the standard message given in DRC to diarrhea patients to the PICHA7 mHealth program. The standard message arm is the standard recommendation given in DRC to diarrhea patients at discharge on the use of oral rehydration solution (ORS) for dehydration, and the importance of handwashing with soap and water treatment for disease prevention. The PICHA7 mHealth program arm will first be delivered during a health facility visit by a health promoter bedside to a diarrhea patient (adults and child) and their accompanying household members during the time of illness followed by two home visits during the 7-day high risk period for diarrheal disease transmission. The health promoter delivers a pictorial WASH module on how diarrhea can spread, and instructions on handwashing with soap, water treatment, and safe water storage. A diarrhea prevention package is provided containing: a one-month supply of chlorine tablets for water treatment, a soapy water bottle for handwashing, a handwashing station, and a water vessel with a lid and tap to ensure safe water storage. After health facility delivery of the program, patient households receive weekly voice and text messages from the PICHA7 mHealth program over 12 months on the recommended WASH behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Diarrhea patients presenting with three or more loose stools over a 24h period
* Having no running water inside of their home
* Plan to reside in Bukavu for the next 12 months
* Have a child <5 years in their household
* Have a working mobile phone in the household

Exclusion Criteria:

* No one will be excluded because of age, sex, religion, or sexual preference
* Presenting at the health facility with a fever (COVID-19 prevention)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2900 (Estimated)
Dates: Start 2021-12-22 (Actual); Primary Completion 2026-12-22 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Diarrhea among household members | 12 months
  Self-reported or caregiver reported diarrhea (3 or more loose stools for a 24 hour period)

SECONDARY OUTCOMES:
Child development for children under 5 years of age | 12 and 24 months after enrollment
  Assessed by Extended Age and Stages Assessment Questionnaire (EASQ)
Handwashing with soap at stool and food related events | 1 week and 1, 3, 6, 9, 12, 18, and 24 months after enrollment
  Rate of patient household members handwashing with soap at stool and food related events measured measured using a 5 hour structured observation tool in the household using our developed forms (George CM, Monira S, Zohura F, Thomas ED, Hasan MT, Parvin T, Hasan K, Rashid MU, Papri N, Islam A, Rahman Z. Effects of a water, sanitation, and hygiene mobile health program on diarrhea and child growth in Bangladesh: a cluster-randomized controlled trial of the cholera hospital-based intervention for 7 days (CHoBI7) mobile health program. Clinical Infectious Diseases. 2021 Nov 1;73(9):e2560-8.)
Free chlorine concentration in stored drinking water | 1 week and 1, 3, 6, 9, 12, 18, and 24 months after enrollment
  mg / Liter
Presence of Vibrio cholerae and E. coli in stored drinking water | 1 week and 1, 3, 6, 9, 12, 18, and 24 months after enrollment
  bacterial culture
WASH psychosocial factors | 1 week and 12 and 24 months after enrollment
  Water, Sanitation, and Hygiene (WASH) psychosocial risk factor questionnaire
non-baseline cholera infections confirmed by bacterial culture among household members of cholera patients | 1 Month
  via rapid dipstick test (RDT) and bacterial culture
Height-for-age among children under 2 years of age | 12 and 24 months after enrollment
  Height and age measurements among children under 2 years of age assessed over a 12-month period were used to calculate height-for-age z-scores according to the World Health Organization child growth standards
Height-for-age among children under 5 years of age | 12 and 24 months after enrollment
  Height and age measurements among children under 5 years of age assessed over a 12-month period were used to calculate height-for-age z-scores according to the World Health Organization child growth standards
Weight-for-age among children under 2 years of age | 12 and 24 months after enrollment
  Weight and age measurements among children under 2 years of age assessed over a 12-month period were used to calculate weight-for-age z-scores according to the World Health Organization child growth standards
Weight-for-age among children under 5 years of age | 12 and 24 months after enrollment
  Weight and age measurements among children under 5 years of age assessed over a 12-month period were used to calculate weight-for-age z-scores according to the World Health Organization child growth standards
Weight-for-height among children under 2 years of age | 12 and 24 months after enrollment
  Height, weight and age measurements among children under 2 years of age assessed over a 12-month period were used to calculate weight-for-height z-scores according to the World Health Organization child growth standards
Weight-for-height among children under 5 years of age | 12 and 24 months after enrollment
  Height, weight and age measurements among children under 5 years of age assessed over a 12-month period were used to calculate weight-for-height z-scores according to the World Health Organization child growth standards
Diarrhea events among household members | 24 months
  Self-reported or caregiver reported diarrhea (3 or more loose stools for a 24 hour period)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Marie George, PhD, Principal Investigator — Associate Professor
Locations (2):
- Democratic Republic of the Congo (2):
  - General Provincial Reference Hospital of Bukavu, Bukavu, South Kivu
  - Université Catholique de Bukavu, Bukavu, South Kivu

IPD SHARING:
Plan to Share IPD: No
All data will be de-identified and available to our collaborators

REFERENCES:
- [Derived] Sanvura P, Endres K, Bisimwa JC, Perin J, Cikomola C, Bengehya J, Maheshe G, Boroto R, Mwishingo A, Bisimwa L, Williams C, George CM. Process evaluation for the delivery of a water, sanitation, and hygiene mobile health program: randomized controlled trial of the WASHmobile PICHA7 program. Trop Med Health. 2026 Jan 7;54(1):15. doi: 10.1186/s41182-025-00881-8. PMID 41501962
- [Derived] George CM, Sanvura P, Bisimwa JC, Endres K, Namunesha A, Felicien W, Banywesize BM, Williams C, Perin J, Sack DA, Boroto R, Nsimire G, Rugusha F, Endeleya F, Kitumaini P, Lunyelunye C, Buhendwa E, Kitumaini Bujiriri P, Tumusifu J, Munyerenkana B, Trivedi S, Davis KL, Jacobson K, Al-Dandashi KM, Leung DT, Caulfield LE, Bengehya J, Maheshe G, Cikomola C, Mwishingo A, Bisimwa L. Effects of a Water, Sanitation, and Hygiene Program on Diarrhea, Cholera, and Child Growth in the Democratic Republic of the Congo: A Cluster-Randomized Controlled Trial of the Preventative Intervention for Cholera for 7 Days (PICHA7 WASHmobile) Mobile Health Program. Clin Infect Dis. 2025 Nov 6;81(4):785-796. doi: 10.1093/cid/ciaf417. PMID 41206550